CLINICAL TRIAL: NCT02026557
Title: Mortality Among Children With Congenital Heart Defects in Norway
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Oslo (Other); University of Bergen (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/392
Record Dates: First submitted 2013-07-02; First posted 2014-01-03 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe mortality among children with congenital heart defects in Norway

ELIGIBILITY:
Inclusion Criteria:

* children with congenital heart defects

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Oslo University hospital´s registry of patients with congenital heart diseases
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 1994-01 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of death until 31 dec 2012 among Norwegian children with congenital heart defects born 1994-2009 | 31.12.2010

CONTACTS AND LOCATIONS:
Overall Officials: Jarle Jortveit, PhD, Principal Investigator — Sorlandet Hospital

REFERENCES:
- [Derived] Jortveit J, Leirgul E, Eskedal L, Greve G, Fomina T, Dohlen G, Tell GS, Birkeland S, Oyen N, Holmstrom H. Mortality and complications in 3495 children with isolated ventricular septal defects. Arch Dis Child. 2016 Sep;101(9):808-13. doi: 10.1136/archdischild-2015-310154. Epub 2016 Apr 18. PMID 27091847